CLINICAL TRIAL: NCT01108679
Title: Neurocognitive Effects of Buprenorphine Among HIV+ and HIV-Opioid Users
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Montefiore Medical Center (Other); Fordham University (Other)
Responsible Party: Principal Investigator, Julia H. Arnsten, Prof., Dept of Medicine, Albert Einstein College of Medicine
Other Study IDs: 2009-471
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Opioid-related Disorders; Buprenorphine; HIV; Cognition; HIV Infections
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | US Export: Yes

GROUPS / COHORTS (1):
- Buprenorphine: Opioid-dependent drug users who are initiating buprenorphine treatment at the Albert Einstein College of Medicine Division of Substance Abuse (DoSA) or at Montefiore's Comprehensive Health Care Center (CHCC).

SUMMARY:
The purpose of this study is to examine how Buprenorphine, a form of opioid addiction treatment, changes the ability to think and reason among people addicted to opiates, who are either HIV negative or HIV positive. In addition, blood samples will be stored for HIV+ and HIV- individuals who take buprenorphine to study its effect. This study hypothesizes that the HIV positive participants will demonstrate significant improvement in thinking and reasoning ability at 3 and 6 months compared to baseline, but that their thinking and reasoning ability will still be lower than HIV negative participants. This study also hypothesizes the biomarkers in participants' blood samples will be associated with measures of change in thinking and reasoning ability.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-serostatus
* English-speaking
* Age 18-60
* Able to give voluntary, signed informed consent
* Plan to initiate buprenorphine treatment in the next month.

Exclusion Criteria:

* Over age 60: Participants over the age of 60 will be excluded, as normal age-associated cognitive changes may confound neuropsychological (NP) assessment and diagnosis of HIV-related cognitive disorders.
* Neurologic: History of head injury with loss of consciousness for greater than 12 hours; previous penetrating skull wounds; previous brain surgery; known seizure disorder, or any other non-HIV related CNS disorders that might affect neurocognitive functioning (e.g., previous cerebrovascular accident, Parkinson's disease, multiple sclerosis, brain tumor).
* Medical: e.g. collagen vascular disorder (e.g. lupus), oxygen requiring chronic pulmonary disease,, or end stage renal disease requiring dialysis.
* Psychiatric: Lifetime diagnosis of schizophrenia or bipolar disorder.
* Less than 6 years of education.
* Acute intoxication due to alcohol or other drugs, as assessed by research staff.
* Use of buprenorphine in the past month, either prescribed or purchased on the street.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects for this study will be drug users with a diagnosis of opioid dependence who are initiating buprenorphine therapy at a DoSA clinic or at the CHCC. The study population is expected to reflect the ethnic composition of the opioid-dependent population in the Bronx. This population is composed of 40% women, and is 24% African-American, 58% Hispanic and 17% Caucasian. Both males and females with opioid dependence who are initiating buprenorphine will be recruited for the proposed study, and, based on our previous studies, we expect to recruit high proportions of women and minorities.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-12-01; Primary Completion 2012-02-01 (Actual); Study Completion 2012-02-01 (Actual)

PRIMARY OUTCOMES:
Global Neurocognitive Function | Months 3 and 6
Neurocognitive functioning in the domains of executive functioning, including decision making, processing speed, verbal memory, attention, and motor functioning | Months 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Julia Arnsten, M.D., M.P.H., Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Fordham University, The Bronx, New York
  - Albert Einstein College of Medicine, The Bronx, New York

REFERENCES:
- [Derived] Scott TM, Rivera Mindt M, Cunningham CO, Arias F, Coulehan K, Mangalonzo A, Olsen P, Arnsten JH. Neuropsychological function is improved among opioid dependent adults who adhere to opiate agonist treatment with buprenorphine-naloxone: a preliminary study. Subst Abuse Treat Prev Policy. 2017 Nov 15;12(1):48. doi: 10.1186/s13011-017-0133-2. PMID 29141650